CLINICAL TRIAL: NCT06969430
Title: A Phase 1/2, First-in-human, Multicenter, Open-label Trial Evaluating the Safety, Tolerability, and Antileukemic Activity of Debio 1562M in Participants With Acute Myeloid Leukemia (AML)
Brief Title: A Study to Assess the Safety, Tolerability, and Antileukemic Activity of Debio 1562M in Participants With Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1562M-101; 2024-519610-32 (Other: EU CT Number); U1111-1315-5913 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 (Dose Escalation): Debio 1562M (Experimental): Participants will receive Debio 1562M intravenously in escalating doses, once in every 3 weeks (Q3W), during each 21-day treatment cycle until progression of disease, unacceptable toxicity, participant's withdrawal, or Investigator's decision, or end of study whichever occurs first.
  Interventions: Drug: Debio 1562M
- Phase 1 (Dose Optimization): Debio 1562M (Experimental): Participants will be randomised 1:1 to receive 1 of the 2 Debio 1562M dose(s) and/or dosing schedule(s) selected based on the results from the Phase 1-Dose escalation for further investigation.
  Participants will be randomized to receive one of the 2 selected doses from Phase 1 (dose escalation) for further investigation and selection of recommended dose (RD) for Phase 2. Participants will receive Debio 1562M intravenously, once in every 3 weeks (Q3W), during each 21-day treatment cycle until progression of disease, unacceptable toxicity, participant's withdrawal, or Investigator's decision, or end of study whichever occurs first.
  Interventions: Drug: Debio 1562M
- Phase 2: Debio 1562M (Experimental): Participants will receive RD of Debio 1562M based on the results from Phase 1-Dose optimization. Participants will receive Debio 1562M intravenously, once in every 3 weeks (Q3W), during each 21-day treatment cycle until progression of disease, unacceptable toxicity, participant's withdrawal, or Investigator's decision, or end of study whichever occurs first.
  Interventions: Drug: Debio 1562M

INTERVENTIONS:
Drug: Debio 1562M — Administered as intravenous (IV) infusion

SUMMARY:
The primary purpose of Phase 1 is to assess the doses studied under Phase 1 (Dose Escalation) Arm A and identify the recommended dose (RD) for further development (Dose optimization).

The primary objective of Phase 2 is to evaluate the antileukemic activity of Debio 1562M.

ELIGIBILITY:
Inclusion Criteria:

* For Phase 1-Dose escalation: Relapsed/refractory (R/R) AML (excluding acute promyelocytic leukemia) based on World Health Organization (WHO) Classification 2022 and relapsed/refractory higher-risk myelodysplastic syndrome (R/R HR -MDS) (includes high- and very high-risk MDS) as confirmed by the Revised International Prognostic Scoring System (IPSS-R) for whom no standard therapy of proven benefit is available.
* For Phase1-Dose optimization and Phase 2: R/R AML (excluding acute promyelocytic leukemia) based on world health organization (WHO) classification 2022 for whom no standard therapy of proven benefit is available.
* Eastern Cooperative Oncology Group performance (ECOG PS) status ≤2.
* Previous treatment-related toxicities must be resolved to ≤Grade 1 (excluding alopecia).
* Individuals with prior autologous or allogeneic bone marrow (BM) transplant are eligible.
* Prior allogeneic transplant must meet the following conditions: the transplant must have been performed more than 120 days before the first administration of Debio 1562M, the participant must not have ≥Grade 1 active graft versus host disease (GvHD) at the time of trial treatment start and must be off all immunosuppression for at least 2 weeks prior to starting treatment with Debio 1562M. Steroid use [equivalent to ≤20 milligrams (mg) prednisone] before and during the trial is allowed as long as this is not being used as post-transplant immunosuppression or graft versus host disease (GVHD) directed therapy.
* Adequate renal and hepatic function defined as:

  1. Estimated glomerular filtration rate (eGFR) ≥60 milliliter per minute (mL/min) based on the chronic kidney disease-Epidemiology Collaboration based on creatinine (CKD-EPIcr) 2021 equation.
  2. Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN).
  3. Serum total bilirubin level ≤1.5× ULN (for participants with Gilbert's syndrome or chronic blood transfusions, total bilirubin ≤3.0× ULN).

Exclusion criteria:

* Any prior exposure to cluster of differentiation (CD) 37 targeting agents.
* Clinically active infection including known active hepatitis B or C, human immunodeficiency virus infection, or cytomegalovirus or any other known concurrent infectious disease that, in the judgment of the Investigator, would make a participant inappropriate for enrollment into this trial (retesting not required).
* Clinically significant cardiac dysfunction within 6 months before enrollment including New York Heart Association Class III or IV heart failure, uncontrolled angina, myocardial infraction, severe uncontrolled ventricular arrhythmias, QT interval corrected for HR according to Fridericia's formula (QTcF) >470 ms.
* Clinically significant and active cardiopulmonary disease.
* Other malignancies, except of:

  1. Hematologic malignancies other than those being investigated for which individuals are not on active antineoplastic therapy
  2. Nonhematologic malignancies in remission and for which individuals must have completed all antineoplastic therapy at least 6 months before trial treatment start and all treatment-related toxicities must have resolved to ≤Grade 1.
* Evidence for active central nervous system (CNS) leukemia involvement. If the participant has a prior history of CNS AML, the participant must have at least 2 negative cerebrospinal fluid (CSF) analyses and either a magnetic resonance imaging (MRI) or computed tomography (CT) (if MRI is not feasible) of the brain demonstrating no evidence of CNS disease.
* Evidence of peripheral neuropathy Grade ≥2.
* History of hypersensitivity to Debio 1562M (including its components), or any of its excipients.
* Treatment with any antileukemic therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic, or any investigational agent within 14 days or within 5 half-lives of the investigational treatment prior to first dose of trial treatment, whichever is shorter. Hydroxyurea may be given prior to and after trial treatment start for control of leukocytosis.
* Major surgery within 4 weeks prior to the start of treatment, or participant who have not recovered from side effects of the surgery.
* Pregnancy or breastfeeding.

Note: Other Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (Dose Escalation): Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) | Up to Day 28
Phase 1: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) | Up to Day 219
Phase 1 (Dose Optimization): Recommended Dose (RD) of Debio 1562M | Up to Day 198

SECONDARY OUTCOMES:
Phases 1 and 2: Overall Response (OR) | Up to Day 198
Phases 1 and 2: Percentage of Participants with CR | Up to Day 198
Phases 1 and 2: Percentage of Participants With CR+ CRh | Up to Day 198
Phases 1 and 2: Percentage of Participants With Composite Complete Remission (cCR) | Up to Day 198
Phases 1 and 2: Percentage of Participants With Allogeneic Hematopoietic Stem Cell Transplant (ASCT) | Up to Day 198
Phases 1 and 2: Change From Baseline in Blood Blast Count | Baseline upto Day 198
Phases 1 and 2: Duration of Remission (DOR) | Up to Day 198
Phases 1 and 2: Relapse Free Survival (RFS) | Up to Day 198
Phase 1 (Dose Optimization) and Phase 2: Event Free Survival (EFS) | Up to Day 198
Phase 1 (Dose Optimization) and Phase 2: Overall Survival (OS) | Up to Day 198
Phases 1 and 2: Plasma Concentration of Debio 1562M and its Metabolites | Pre-dose and at multiple time points up to Day 198
Phase 1 (Dose Optimization) and Phase 2: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) | Up to Day 219

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Moffitt Cancer Center and Research Institute Hospital, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - START Midwest, Grand Rapids, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - The Ohio Sate University, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No